CLINICAL TRIAL: NCT01913457
Title: Evaluation of Lung Doppler Signals in Pediatric and Adult Patients
Brief Title: Measurements and Characterization of Doppler Signals From the Right Chest in Pediatric and Adult Patients
Status: Terminated | Type: Observational
Sponsor: Echosense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DOP018/25388
Record Dates: First submitted 2013-07-25; First posted 2013-08-01 (Estimated); Last update posted 2022-03-23 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Hypertension
Keywords: Ultrasound Doppler; Lungs; Pulmonary artery hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Adults w/ PH: Subjects above 18y scheduled to undergo RHC for Doppler ultrasound external right chest wall tests
  Interventions: Radiation: Ultrasound Doppler
- Children w/ PH: Children 0-18y old scheduled to RHC
  Interventions: Radiation: Ultrasound Doppler
- Children control: Children 0-18y old w/o PH for Lung Doppler tests as controls
  Interventions: Radiation: Ultrasound Doppler

INTERVENTIONS:
Radiation: Ultrasound Doppler — Doppler Ultrasound recording on external right chest wall

SUMMARY:
Recently it has been shown that clear reproducible Doppler signals can be recorded from the lung parenchyma by means of a pulsed Doppler ultrasound system incorporating a special signal processing package parametric Doppler, TPD, EchoSense Ltd., Haifa, Israel). These lung Doppler signals (LDS) are in full synchrony with the cardiac cycle and can be obtained from the lungs, including areas remote from the heart and main pulmonary vessels. The LDS waves typically have peak velocities of up to 30 cm/s and are of relatively high power, making it possible to detect them despite the aforementioned attenuation by the air in the lungs. The LDS are thought to represent the radial wall movement of small pulmonary blood vessels, caused by pressure pulse waves of cardiac origin which propagate throughout the lung vasculature. The LDS may contain information of significant diagnostic and physiological value regarding the pulmonary parenchyma and vasculature, as well as the cardio-vascular system in general.

Pulmonary arterial hypertension (PAH) is a condition characterized by reshaping of the small pulmonary arteries with increase in pulmonary vascular resistance, leading gradually to right-sided cardiac failure. A trans-thoracic echocardiograph (TTE) is a test classically undertaken in order to screen for pulmonary hypertension. However, the systolic pulmonary artery pressure (SPAP) values thereby obtained are often imprecise and depend upon the expertise of the individual carrying out the test. Therefore, the pulmonary arterial pressure and cardiac output values have to be ascertained with a right-sided cardiac catheterization, which is considered the gold-standard, but is invasive.

In a pilot study of adult PAH patients (unpublished), lung Doppler signals have been shown to have the potential to diagnose pulmonary hypertension in two different ways: First, by measuring the degree of attenuation of the LDS during acute pressure rise in the chest cavity (i.e. during Valsalva maneuver). Second, by detecting differences between the LDS in patients with PAH and control subjects.

One of the objectives of the present study is to evaluate the lung Doppler signals in pediatric patients of various age groups, with and without pulmonary vascular disease. The second objective of the study is to verify previous findings of abnormal lung Doppler signals in adult patients with pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing RHC:
* Males or females aged over 18 years
* With suspicion or diagnosis of pulmonary hypertension.
* Scheduled to undergo right heart catheterization
* Able and willing to give informed consent

Pediatric patients undergoing RHC:

* Males or females aged 0-18 years
* Scheduled to undergo right hear catheterization
* Parents willing to give informed consent

Pediatric patients without significant cardio-pulmonary diseases:

* Males or females aged 0-18 years Not known to have a significant cardiac or pulmonary disease
* Legal guardians willing to give informed consent

Exclusion Criteria:

* -Hemodynamically unstable patients.
* For adult and pediatric patients undergoing right heart catheterization:

  a. Any contra-indication to perform the procedure
* For adults only:

  1. Patients incapable of performing a Valsalva maneuver
  2. Patients with recent (within the past 3 months) myocardial infarction, high degree AV block, severe aortic stenosis or open angle glaucoma

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study targets to enroll 200 patients (see inclusion criteria): 100 patients will be children without cardiopulmonary diseases, 50 patients will be children undergoing heart catheterization, 50 patients will be adults undergoing heart catheterization
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Diagnose specific pattern of LDS in children by features as velocity & power in comparison to adult LDS pattern. | 1 year to collect all data and obtain an average diagnostic pattern

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Feinstein, MD, Principal Investigator — Stanford Hospital and Clinics and Lucile Packard Children's Hospital
Locations (2):
- United States (2):
  - Stanford Hospital and Clinics and Lucile Packard Children's Hospital, Palo Alto, California
  - Stanford university hospital, Palo Alto, California